CLINICAL TRIAL: NCT02390336
Title: The Immediate Effects of Mulligan Mobilization With Movement Technique in Pain, Range of Motion and Physical Function in Patients With Osteoarthritis of the Hip
Brief Title: Mobilization With Movement in Patients With Osteoarthritis of the Hip
Acronym: MWM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natália Maria Oliveira Campelo (Other)
Responsible Party: Sponsor-Investigator, Natália Maria Oliveira Campelo, Profesor, Escola Superior de Tecnologia da Saúde do Porto
Organization: Escola Superior de Tecnologia da Saúde do Porto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NC-002
Record Dates: First submitted 2015-03-03; First posted 2015-03-17 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis Hip; Joint Disease; Musculoskeletal Diseases; Pathologic Processes
Keywords: Osteoarthritis of the hip; Pain; Range of Motion; Physical Function; Manual Therapy
MeSH Terms: conditions — Osteoarthritis, Hip; Joint Diseases; Musculoskeletal Diseases; Pathologic Processes; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real mobilization-with-movement (MWM) (Experimental): In each volunteer of this group, the blind assessor will perform the pre-intervention measurements of intensity of pain, range of motion and physical function tests.
  Next, the therapist will performed the real mobilization-with-movement. Then, all measurements, before described, will be repeated, by the assessor.
  Interventions: Other: Real mobilization-with-movement (MWM)
- Sham mobilization-with-movement (MWM) (Sham Comparator): In each volunteer of this group, the blind assessor will perform the pre-intervention measurements of intensity of pain, range of motion and physical function tests.
  Next, the therapist will performed the sham mobilization-with-movement. Then, all measurements, before described, will be repeated, by the assessor.
  Interventions: Other: Sham mobilization-with-movement (MWM)

INTERVENTIONS:
Other: Real mobilization-with-movement (MWM) — For the MWM group, the investigator applied two techniques of mobilization with movement: one for flexion and one for medial rotation of the hip. With the hip in flexion, a stabilizing belt was placed on the medial side of the participant's thigh closest to the joint interline. The belt was placed around the pelvic region of the physical therapist, keeping a perpendicular direction to the participant's thigh. Maintaining a side slip, it was carried out a passive movement of 1) hip flexion (3x10) and 2) medial hip rotation (3x10) by the physiotherapist throughout painless amplitude.
  Other Names: Group Experimental: mobilization-with-movement (MWM)
  Arms: Real mobilization-with-movement (MWM)
Other: Sham mobilization-with-movement (MWM) — In the sham group, the investigators conducted a technical simulation. The positioning of the patient and the physical therapist was the same, however, no accessory mobilization was performed with the help of the belt and did not performed repeated movements of passive flexion or medial rotation.
  Other Names: Group Sham: mobilization-with-movement (MWM)
  Arms: Sham mobilization-with-movement (MWM)

SUMMARY:
The concept of mobilization with movement, also referred to as a Mulligan mobilization, has not been studied in patients with hip osteoarthritis, subsisting questions about the possible effects in this population. The aim of this randomized controlled study is to compare the immediate effects of Mulligan mobilization with movement technique of pain, range of motion and physical function in patients with osteoarthritis of the hip.

DETAILED DESCRIPTION:
Mulligan original theory for the efficacy of a Mobilization With Movement (MWM) is based on the concept associated with a "positional joint failure," which occurs due to injury and may lead to a change in the joint alignment and hence its biomechanical resulting in symptoms such as pain, joint stiffness or weakness. To perform the MWM technique it is required to implement many criteria. During execution is applied an maintained accessory glide in order to correct the positional fault, while a physiological movement or action that usually caused the pain is performed actively or passively. A key component for the MWM is that pain should always be reduced and / or eliminated during application.

All study participants will be submitted to an initial assessment protocol to determine the intensity of pain, the range of motion (ROM) in flexion and internal rotation of the hip and the collection of physical function parameters. After that, the intervention will be performed for each group, and then the re-evaluation will be carried out (final evaluation), pain intensity, ROM and physical function tests..

ELIGIBILITY:
Inclusion Criteria:

clinical criteria for the diagnosis of osteoarthritis of the hip (sensitivity 86% and specificity 75%) are:

* Medial hip rotation ≥15º, pain during medial rotation of the hip, morning fatigue in hip> 60 minutes and older than 50 years or
* Medial hip rotation <15, hip flexion ≤ 115

Exclusion Criteria:

* Previous surgery or hip replacement or knee joint
* Another surgery in the lower extremities performed within 6 months, rheumatoid arthritis
* Uncontrolled hypertension or risk (moderate - high) of cardiac complications during exercise
* Disability unrelated to the hip or knee to prevent the safe participation during exercise, appliance of manual therapy or during march: vision problems affecting mobility, body weight equal to or greater than 155 kg, primary neurogenic disorder or significantly limitation of the lumbar level,advanced osteoporosis with manual therapy or other treatment technique that may interfere with the study
* With inability to understand the instructions and complete the study assessments

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in the intensity of hip pain before and after the treatment | participants will be assessed before and after intervention (interval: 15-20 minutes)
  Participants were asked to rate the intensity of their pain using an 11-point numerical pain rating scale (NPRS; 0: no pain; 10: maximum pain).

SECONDARY OUTCOMES:
Changes in the range of motion for the hip flexion before and after the treatment | participants will be assessed before and after intervention (interval: 15-20 minutes)
  Assess ROM of the hip joint was used a universal goniometer BIOMET® (CAT.No.567330), it was considered a valid instrument to measure hip flexion.
Changes in the range of motion for the medial hip rotation before and after the treatment | participants will be assessed before and after intervention (interval: 15-20 minutes)
  Assess ROM of the hip joint was used a universal goniometer BIOMET® (CAT.No.567330), it was considered a valid instrument to measure medial hip rotation.
Changes in the performing time of the physical function test timed up and go before and after the treatment | participants will be assessed before and after intervention (interval: 15-20 minutes)
  The Timed "Up and Go" Test (TUG) is presented as a test that simulates some functional maneuvers of daily life, like, getting up, walking, running laps and siting down.
Changes in the repetitions of the physical function test 30 seg sit to stand before and after the treatment | participants will be assessed before and after intervention (interval: 15-20 minutes)
  The 30 sec Sit to Stand test or 30 sec Chair Stand Test (CST) is the functional evaluation of the strength of the lower limbs.Is to repeat the activity of sit and lift a maximum number of times during 30 seconds.
Changes in the performing time of the physical function test 40 m. self placed walk before and after the treatment | participants will be assessed before and after intervention (interval: 15-20 minutes)
  The test 40m Self Placed Walk (SPWT) consists is the functional assessment of physical ability of an individual coursing short distances (40 meters).

CONTACTS AND LOCATIONS:
Overall Officials: Natália Campelo, PhD, Study Director — Polytechnic Institute of Porto (Portugal); Francisco Neto, MSc, Study Director — Polytechnic Institute of Porto (Portugal); Carlos Beselga, MSc, Principal Investigator — Polytechnic Institute of Porto (Portugal); Francisco A Sendín, PhD, Study Director — University of Salamanca (Spain)

REFERENCES:
- [Background] Vicenzino B, Paungmali A, Teys P. Mulligan's mobilization-with-movement, positional faults and pain relief: current concepts from a critical review of literature. Man Ther. 2007 May;12(2):98-108. doi: 10.1016/j.math.2006.07.012. Epub 2006 Sep 7. PMID 16959529
- [Background] Hoeksma HL, Dekker J, Ronday HK, Breedveld FC, Van den Ende CH. Manual therapy in osteoarthritis of the hip: outcome in subgroups of patients. Rheumatology (Oxford). 2005 Apr;44(4):461-4. doi: 10.1093/rheumatology/keh482. Epub 2005 Feb 3. PMID 15695307
- [Background] Botha-Scheepers S, Riyazi N, Kroon HM, Scharloo M, Houwing-Duistermaat JJ, Slagboom E, Rosendaal FR, Breedveld FC, Kloppenburg M. Activity limitations in the lower extremities in patients with osteoarthritis: the modifying effects of illness perceptions and mental health. Osteoarthritis Cartilage. 2006 Nov;14(11):1104-10. doi: 10.1016/j.joca.2006.04.011. Epub 2006 Jun 5. PMID 16740397
- [Background] French HP, Cusack T, Brennan A, Caffrey A, Conroy R, Cuddy V, FitzGerald OM, Fitzpatrick M, Gilsenan C, Kane D, O'Connell PG, White B, McCarthy GM. Exercise and manual physiotherapy arthritis research trial (EMPART) for osteoarthritis of the hip: a multicenter randomized controlled trial. Arch Phys Med Rehabil. 2013 Feb;94(2):302-14. doi: 10.1016/j.apmr.2012.09.030. Epub 2012 Oct 16. PMID 23084955
- [Background] Hando BR, Gill NW, Walker MJ, Garber M. Short- and long-term clinical outcomes following a standardized protocol of orthopedic manual physical therapy and exercise in individuals with osteoarthritis of the hip: a case series. J Man Manip Ther. 2012 Nov;20(4):192-200. doi: 10.1179/2042618612Y.0000000013. PMID 24179327
- [Derived] Beselga C, Neto F, Alburquerque-Sendin F, Hall T, Oliveira-Campelo N. Immediate effects of hip mobilization with movement in patients with hip osteoarthritis: A randomised controlled trial. Man Ther. 2016 Apr;22:80-5. doi: 10.1016/j.math.2015.10.007. Epub 2015 Oct 31. PMID 26559319